CLINICAL TRIAL: NCT00000789
Title: A Randomized, Comparative Trial of Zidovudine (AZT) Versus 2',3'-Didehydro-3'-Deoxythymidine (Stavudine; d4T) in Children With HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 240; 11217 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Stavudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Stavudine; Zidovudine

INTERVENTIONS:
Drug: Stavudine
Drug: Zidovudine

SUMMARY:
PRIMARY: To compare the relative safety and tolerance of oral zidovudine (AZT) versus oral stavudine (d4T) in symptomatic HIV-infected children.

SECONDARY: To compare the clinical, virologic, and immunologic responses between the two treatment groups, and to obtain pharmacokinetic data for both drugs.

At present, AZT is considered the drug of choice for initial treatment of most children with HIV infection, although disease progression or drug intolerance is associated with its long-term use. In preliminary studies in children, d4T, another HIV inhibitor, has been well tolerated, although an optimum dose has not been determined.

DETAILED DESCRIPTION:
At present, AZT is considered the drug of choice for initial treatment of most children with HIV infection, although disease progression or drug intolerance is associated with its long-term use. In preliminary studies in children, d4T, another HIV inhibitor, has been well tolerated, although an optimum dose has not been determined.

Patients are randomized to receive either oral AZT or oral d4T. Treatment continues until the last patient enrolled has received 52 weeks of therapy, or until the study is terminated.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Recommended:

* PCP prophylaxis.

Allowed:

* Immunoglobulin.
* Erythropoietin, G-CSF, and GM-CSF.
* Corticosteroids.
* Ethionamide or isoniazid for TB if no alternative is available.
* Pyridoxine (up to 50 mg/day) as vitamin supplement.

Patients must have:

* Symptomatic HIV infection.
* No more than 6 weeks of prior antiretroviral or immunomodulator therapy (other than steroids and IVIG).
* Consent of parent or guardian.

NOTE:

* Coenrollment on another ACTG protocol not involving antiretroviral therapy is permitted.

Prior Medication:

Allowed:

* Maternal immunomodulator or antiretroviral therapy (including during pregnancy).
* Antiretroviral therapy prior to 2 months.
* Up to 6 weeks of prior antiretroviral therapy or specific immunomodulator therapy (other than corticosteroids and IVIG).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Current grade 3 or worse neuropathy / lower motor neuropathy.
* Other grade 3 or worse clinical or laboratory toxicities.
* Known intolerance to either AZT or d4T.

Concurrent Medication:

Excluded:

* Chemotherapy for active malignancy.

Patients with the following prior conditions are excluded:

* History of grade 3 or worse neuropathy/lower motor neuropathy.

Prior Medication:

Excluded:

* More than 6 weeks of prior antiretroviral or immunomodulator therapy.
* Antiretroviral or immunomodulator therapy within 7 days prior to study entry. Ongoing drug or alcohol abuse.

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230
Dates: Study Completion 1998-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kline M, Study Chair; Van Dyke R, Study Chair
Locations (54):
- United States (51):
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Usc La Nichd Crs, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Univ. of Connecticut Health Ctr., Dept. of Ped., Farmington, Connecticut
  - Yale Univ. School of Medicine - Dept. of Peds., Div. of Infectious Disease, New Haven, Connecticut
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Emory Univ. School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Atlanta, Georgia
  - Cook County Hosp., Chicago, Illinois
  - Univ. of Illinois College of Medicine at Chicago, Dept. of Peds., Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - Cooper Univ. Hosp., Camden, New Jersey
  - UMDNJ - Robert Wood Johnson, New Brunswick, New Jersey
  - St. Joseph's Hosp. & Med. Ctr. of New Jersey, Paterson, New Jersey
  - Children's Hospital at Albany Medical Center, Dept. of Peds., Albany, New York
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - North Shore-Long Island Jewish Health System, Dept. of Peds., Great Neck, New York
  - Schneider Children's Hosp., Div. of Infectious Diseases, New Hyde Park, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Metropolitan Hosp. NICHD CRS, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Incarnation Children's Ctr., New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - UNC at Chapel Hill School of Medicine - Dept. of Peds., Div. of Immunology & Infectious Diseases, Chapel Hill, North Carolina
  - DUMC Ped. CRS, Durham, North Carolina
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
  - Med. Univ. of South Carolina, Div. of Ped. Infectious Diseases, Charleston, South Carolina
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Children's Med. Ctr. Dallas, Dallas, Texas
  - Texas Children's Hosp. CRS, Houston, Texas
  - UW School of Medicine - CHRMC, Seattle, Washington
- Puerto Rico (3):
  - Univ. Hosp. Ramón Ruiz Arnau, Dept. of Peds., Bayamón
  - San Juan City Hosp. PR NICHD CRS, San Juan
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan

REFERENCES:
- [Background] Kline MW, Fletcher CV, Federici ME, Harris AT, Evans KD, Rutkiewicz VL, Shearer WT, Dunkle LM. Combination therapy with stavudine and didanosine in children with advanced human immunodeficiency virus infection: pharmacokinetic properties, safety, and immunologic and virologic effects. Pediatrics. 1996 Jun;97(6 Pt 1):886-90. PMID 8657531
- [Background] McKinney RE Jr. Ongoing and future trials of antiretroviral therapy in the pediatric AIDS clinical trials group (PACTG). Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:173
- [Background] Kline MW, Van Dyke RB, Lindsey JC, Gwynne M, Culnane M, McKinney RE Jr, Nichols S, Mitchell WG, Yogev R, Hutcheon N. A randomized comparative trial of stavudine (d4T) versus zidovudine (ZDV, AZT) in children with human immunodeficiency virus infection. AIDS Clinical Trials Group 240 Team. Pediatrics. 1998 Feb;101(2):214-20. doi: 10.1542/peds.101.2.214. PMID 9445494
- [Background] Perrier M, Schwarz T, Gonzalez O, Brounts S. Squamous cell carcinoma invading the right temporomandibular joint in a Belgian mare. Can Vet J. 2010 Aug;51(8):885-7. PMID 21037891